CLINICAL TRIAL: NCT04849481
Title: The Research Plan of Taiwan Precision Medicine: Lung Cancer
Brief Title: The Research Plan of Taiwan Precision Medicine
Status: Recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: T1521
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Non-small-cell Lung Cancer
Keywords: non-small-cell lung cancer, next-generation sequencing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Next-generation sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-small-cell lung cancer (NSCLC) is one of the top three most common cancers in Taiwan. Targetable driver mutations in NSCLC are more prevalent in Asian population compared to those in Western population, which offers chances to apply suitable targeted therapies worldwide. For patients who failed to the treatment of tyrosine kinase inhibitors (TKIs), the genetic mutations from next-generation sequencing (NGS) reports can serve as the reference of treatment selection. Moreover, the expression of PD-1/PD-L1 serves as a helpful indicator for the response of immune checkpoint inhibitors (ICIs). On the other hand, patients with wild-type EGFR/ALK mutations and PD-L1-negative NSCLC who received chemotherapy had relative poorer survival than those received suitable targeted therapies and ICIs. To further elucidate the underlying molecular genomic aberrations, as well as the clinical demographics and therapeutic outcomes in above subpopulations, it is necessary to have a national, multi-centers and population-focused research project to collect data completely. Tumor tissue will be collected from advanced NSCLC patients with wild-type EGFR/ALK or with EGFR/ALK mutation after resistant to TKIs for next-generation sequencing analysis in a platform of data storage and sharing. The purpose of the precision medicine project is to establish tumor molecular profiling of specific NSCLC populations in Taiwan, to facilitate patients to have corresponding potential targeted therapeutics and suitable clinical trials, and to extend the median overall survival.

DETAILED DESCRIPTION:
Development of an integrated database of genetic background from treatment-naïve and TKI-refractory populations, clinical information, and therapeutic outcomes in advanced NSCLC.

1. To enroll 550 patients who fit the criteria of this study in the enrolled period.
2. To perform large-scale NGS analysis for specific populations, to create a map containing important genetic characteristics to help understand the mechanisms of drug resistance, and to find novel treatment strategies.
3. To collect tumor sample for NGS testing
4. To record previous therapeutic agents and accompanying treatment response and adverse events

ELIGIBILITY:
Inclusion Criteria

1. Ages 20 and above.
2. Pathological reports showed adenocarcinoma, squamous cell carcinoma, large cell carcinoma, adenosquamous carcinoma, and sacromatoid carcinoma.
3. For patients with squamous cell carcinoma, only never smokers and light smokers (less than 10 cigarettes per day) are indicated.
4. For patients with advanced EGFR (-) and ALK (-) adenocarcinoma or other histological types regardless of EGFR/ALK status, treatment-naïve or failure to ≤ two lines of systemic treatment is allowed.
5. For patients with advanced EGFR (+) or ALK (+) adenocarcinoma, failure to ≤ two lines of systemic treatment, including tyrosine kinase inhibitor is allowed.
6. For patients with advanced EGFR exon 20 insertion/mutation (excluding T790M mutation) adenocarcinoma, failure to ≤ four lines of systemic treatment, including tyrosine kinase inhibitor is allowed.
7. Reacquisition of tumor tissue after the failure of previous systemic treatment
8. Willingness to provide the residual biopsy/operative slides.
9. Life expectancy more than 3 months.
10. Patients fully understand the protocol with the willingness to have regular follow-up.
11. For patients with advanced EGFR exon 20 insertion/mutation (excluding T790M mutation) adenocarcinoma: if the patient had died before 2022/07/31, the waiver of Informed Consent Form(s) is allowed under the permission of Independent Ethics Committee/Institutional Review Board (IEC/IRB). Exclusion Criteria

1.Inability to cooperate by providing a complete medical history. 2.No available tumor tissues for genetic testing. 3.Undesirable compliance.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. For patients with advanced EGFR/ALK (-) tumors, treatment-naïve or failure to ≤ two lines of systemic treatment.
  2. For patients with advanced EGFR/ALK (+) tumors, failure to ≤ two lines of systemic treatment, such as tyrosine kinase inhibitors.
  3. patients with advanced EGFR exon 20 insertion/mutation (excluding T790M mutation) adenocarcinoma, failure to ≤ four lines of systemic treatment, including tyrosine kinase inhibitor is allowed.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To perform large-scale NGS analysis for specific populations, create a map containing important genetic characteristics to help understand the mechanisms of drug resistance, and find novel treatment strategies. | 2021/05~2030/12
  Development of an integrated database of genetic background from treatment-naïve and TKI-refractory populations, clinical information, and therapeutic outcomes in advanced NSCLC.

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Jung Chiang, Principal Investigator — National Health Research Institutes, Taiwan
Locations (13):
- Taiwan (13):
  - Chang Gung Medical Foundation, Chiayi City
  - Dalin Tzu Chi Hospital, Dalin
  - Chang Gung Medical Foundation, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taoyuan General Hospital, Taoyuan District